CLINICAL TRIAL: NCT05365399
Title: Evaluation of a Smartphone-based Screening Tool for Neonatal Jaundice in a Ugandan Population
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data collection protocol was not followed-up properly. Results are not reliable
Sponsor: Picterus AS (Industry)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IS 145
Record Dates: First submitted 2022-04-28; First posted 2022-05-09 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Neonatal Jaundice
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enable high qualitative estimation of bilirubin levels in the blood of new-borns (Other): In this study we aim to collect data of newborns with wider range of bilirubin levels and high melanin content, and additionally measurements of skin color reflectance with a spectrophotometer, to adjust the Picterus JP algorithm and optimize the app performance. This will enable a high qualitative estimation of bilirubin levels in the blood of new-borns for all skin colors. .
  Interventions: Device: smartphone-based screening tool for neonatal jaundice

INTERVENTIONS:
Device: smartphone-based screening tool for neonatal jaundice — In this study we aim to collect data of newborns with wider range of bilirubin levels and high melanin content, and additionally measurements of skin color reflectance with a spectrophotometer, to adjust the Picterus JP algorithm and optimize the app performance. This will enable a high qualitative estimation of bilirubin levels in the blood of new-borns for all skin colors. .

SUMMARY:
The general objective of this study is to evaluate the accuracy of a novel smartphone application that estimates bilirubin levels in newborns at HICH Mbarara.

DETAILED DESCRIPTION:
The general objective of this study is to evaluate the accuracy of a novel smartphone application that estimates bilirubin levels in newborns at HICH Mbarara.

The specific objectives for this study are:

To evaluate the correlation between bilirubin estimates from a smartphone application and bilirubin measurements in serum in newborns with varying degree of jaundice To evaluate the correlation between bilirubin estimates from a smartphone application and bilirubin estimates from a standard transcutaneous device in newborns with varying degree of jaundice To evaluate the correlation between bilirubin estimates from a smartphone application and bilirubin estimates from visual inspection in newborns with varying degree of jaundice

ELIGIBILITY:
Inclusion Criteria:

* Infants born with gestational age ≥37 weeks
* Birth weight ≥2000g and ≤4500g
* Age 1 - 14 days
* Infants requiring a blood sample (newborn screening / clinically suspected jaundice)

Exclusion Criteria:

* Infants transferred to the paediatric ward for advanced treatment.
* Infants with a skin rash or other disease that affects the skin where measurements are performed.
* Infants that receive or have received phototherapy in the last 24 hours.
* Infants with an inborn disease

Ages: 24 Hours to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Smartphone application sensitivity (bilirubin levels on newborns) | 5 minutes
  Enable high qualitative estimation of bilirubin levels in the blood of newborns, independent of skin color, using Picterus JP.

SECONDARY OUTCOMES:
Smartphone application sensitivity (bilirubin levels on newborns with high melanin content) in the skin. | 5 minutes
  Enable high qualitative estimation of bilirubin levels in the blood of newborns, independent of skin color, using Picterus JP. Adapt the current algorithm of Picterus JP to newborns with high melanin content in the skin

CONTACTS AND LOCATIONS:
Locations (1):
- Mengo Hospital, Kampala, Uganda